CLINICAL TRIAL: NCT03912610
Title: Study on Brain Structure and Function of Patients With Pain-related Emotion Disorder Via Multi-mode Magnetic Resonance Imaging
Brief Title: Study on Brain Structure and Function of Pain-related Emotion Disorder
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhoujie (Other)
Responsible Party: Sponsor-Investigator, Zhoujie, The officer of Science and Education Division, The Third Affiliated hospital of Zhejiang Chinese Medical University
Organization: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Other Study IDs: 2019-01
Record Dates: First submitted 2019-04-04; First posted 2019-04-11 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Osteoarthritis, Knee; Depressive Symptoms; Anxiety State
Keywords: Osteoarthritis of knee; Depressive Symptoms; Anxiety State; Brain Structure and Function; Multi-mode Magnetic Resonance Imaging
MeSH Terms: conditions — Osteoarthritis, Knee; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Health control group: 5 health volunteer are included in the group. Each volunteer will take the functional magnetic resonance examination one to collect the data.
  Interventions: Diagnostic Test: Functional magnetic resonance examination
- Knee osteoarthritis group: 5 patients of knee osteoarthritis accompanied with depression or anxiety are included in the group. Each volunteer will take the functional magnetic resonance examination one to collect the data.
  Interventions: Diagnostic Test: Functional magnetic resonance examination

INTERVENTIONS:
Diagnostic Test: Functional magnetic resonance examination — Functional magnetic resonance examination by a Ultra high field magnetic resonance instrument named MAGNATOM 7T.

SUMMARY:
By the method of multi-mode Magnetic Resonance Imaging, 5 patients with knee osteoarthritis are selected in this trial to observe the possible differences in the brain structure and function from the 5 healthy volunteers.

DETAILED DESCRIPTION:
In this study, 5 patients with knee osteoarthritis and 5 healthy volunteers were selected. The degree of pain is evaluated via visual analogue pain scale (VAS). The emotional state is evaluated by Hamilton anxiety scale (HAMA) or Hamilton depression scale (HAMD). The patients and healthy volunteers who meet the include criteria are include in the research. Then the spontaneous brain electrical activity is collected by multimodal brain magnetic resonance imaging technology. The spontaneous brain electrical activity is analyzed to find the differences between knee osteoarthritis patients and healthy volunteers. Further analysis of resting brain functional connectivity and information exchange changes in multifunctional areas, in order to elaborate the central mechanism of pain and emotion modulation.

ELIGIBILITY:
Inclusion Criteria:

The experimental group was selected as:

* Meet the above diagnostic criteria.
* VAS scale score > 4 points.
* HAMA score > 14 or HAMD score > 17 points.
* Agree to participate in the survey and submit an informed consent form.

The control group was selected as:

* Healthy volunteers who exclude knee osteoarthritis.
* VAS scale score ≤ 4 points.
* HAMA score ≤14 or HAMD score ≤ 17 points.
* Agree to participate in the survey and submit an informed consent form

Exclusion Criteria:

* Rheumatoid arthritis, psoriatic arthritis, gouty arthritis, bone erosion, bone tuberculosis, bone tumor patients.
* Clear diagnosis of traumatic meniscus, cruciate ligament, collateral ligament injury history and patients with history of knee trauma in the past six months.
* Have a heavier heart, brain and other medical conditions and poor overall health.
* In pregnancy, pregnancy or lactation.
* Taking antidepressant and anxiety drugs.
* Participated in other clinical studies within 2 months prior to the start of the study.
* The patient or his licensor is unwilling to sign a written informed consent or is unwilling to follow the research protocol.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study is a single-center randomized controlled clinical trial. It is expected to enroll 5 patients with knee osteoarthritis in the third affiliated hospital of zhejiang university of traditional Chinese medicine and recruit 5 healthy volunteers at the same time.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
blood-oxygen-level dependent (BOLD) signal | the data will be collected the second day when entering group
  BOLD is used in functional magnetic resonance imaging (fMRI) to observe different areas of the brain or other organs, which are found to be active at any given time. The hemoglobin content, blood flow volume and oxygen consumption of special brain regions will be observed via BOLD. Oxyhemoglobin ratio is used in this measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Yuanyuan Wu, Master, Principal Investigator — the Third affilliated Hospital of Zhejiang Chinese Medicine University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tang S, Lu L, Zhang L, Hu X, Bu X, Li H, Hu X, Gao Y, Zeng Z, Gong Q, Huang X. Abnormal amygdala resting-state functional connectivity in adults and adolescents with major depressive disorder: A comparative meta-analysis. EBioMedicine. 2018 Oct;36:436-445. doi: 10.1016/j.ebiom.2018.09.010. Epub 2018 Oct 11. PMID 30316866
- [Background] Ye J, Shen Z, Xu X, Yang S, Chen W, Liu X, Lu Y, Liu F, Lu J, Li N, Sun X, Cheng Y. Abnormal functional connectivity of the amygdala in first-episode and untreated adult major depressive disorder patients with different ages of onset. Neuroreport. 2017 Mar 1;28(4):214-221. doi: 10.1097/WNR.0000000000000733. PMID 28118287
- [Background] Spati J, Hanggi J, Doerig N, Ernst J, Sambataro F, Brakowski J, Jancke L, grosse Holtforth M, Seifritz E, Spinelli S. Prefrontal thinning affects functional connectivity and regional homogeneity of the anterior cingulate cortex in depression. Neuropsychopharmacology. 2015 Jun;40(7):1640-8. doi: 10.1038/npp.2015.8. Epub 2015 Jan 19. PMID 25598428